CLINICAL TRIAL: NCT01751893
Title: A Randomized Double-blind, Placebo-controlled Study of the Effects of Lawsonia Inermis on Palmar-Plantar Erythrodysesthesia Induced by Capecitabine and/or Pegylated Liposomal Doxorubicin
Brief Title: Testing the Effectiveness of Henna on Managing PPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Associate Professor of Oncology and Palliative Care, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AC-PPEHP-88
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Palmar-plantar Erythrodysesthesia (PPE)
Keywords: Hand-foot syndrome; palmar-plantar erythrodysesthesia; capecitabine; pegylated liposomal doxorubicin; henna
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — lawsone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Henna arm (Experimental): Based on the treatment protocol for this study the patients will receive the henna treatment for 4 weeks (supervised treatment for first week and then unsupervised sessions twice a week). The treatment will include the application of the henna mixture (paste) (40gr natural henna and 40ml of purified water) to the affected areas (feet or/and hands) and wear socks or/and gloves. The treatment session will last for 1 hour and then the mixture will be rinsed with fresh water.
  Interventions: Drug: Henna
- Placebo (Placebo Comparator): Based on the treatment protocol for this study the patients in this arm will receive the henna placebo treatment for 4 weeks (supervised treatment for first week and then unsupervised sessions twice a week). The treatment will include the application of the henna placebo mixture (paste) (40gr placebo henna and 40ml of purified water) to the affected areas (feet or/and hands) and wear socks or/and gloves. The treatment session will last for 1 hours and then the mixture will be rinsed with fresh water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Henna — natural henna in the form of paste
  Arms: Henna arm
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The palmar-plantar erythrodysesthesia (PPE) is the only clinical adverse event that commonly occurs with capecitabine and/or pegylated liposomal doxorubicin treatment and it warrants special attention because it is the most common dose-limiting toxicity. this study is designed to test the effectiveness of a henna treatment protocol in the management of capecitabine and/or pegylated liposomal doxorubicin induced palmar-plantar erythrodysesthesia.

DETAILED DESCRIPTION:
This will be a randomized double-blind, placebo-controlled study with 80 cancer patients that will receive chemotherapy treatment with capecitabine and/or pegylated liposomal doxorubicin. The selection of potential participants will be based on pre-determined inclusion and exclusion criteria. Patients will be randomly allocated either to the treatment group or the placebo group. Treatment will be delivered twice a week and assessments will take place at 2, 3, 4, 5 and 6 weeks.

The intervention group will receive the application of henna to the hands and/or feet of the patients and the control group will receive the placebo.

At both baseline and follow-up, patients in both groups will be assessed for their degree of palmar-plantar erythrodysesthesia, the Quality of Life, the need for dose-limiting due to PPE and Pain intensity using standardized rating scales. Data will be analysed with inferential and descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Adult cancer patients (>18)
* Patients receiving capecitabine and/or PLD as monotherapy or in combination with other agents
* Patients that will experience PPE grade 1 or above
* Willing to participate
* Ability to complete the psychometric assessments.
* A performance status of two or less on the Eastern Cooperative Oncology Group (ECOG)

Exclusion Criteria:

* Patients with hypersensitivity to natural henna.
* Patients with pre-existing dermatological condition affecting the hands or feet that may limit the interpretation of results
* Patients on Pyridoxine or nicotine patches
* Patients with a previous history of PPE
* Patients whose chemotherapy was discontinued for more than a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline PPE Grade at 3,4, 5,6 weeks | 3, 4, 5 and 6 weeks
  The grade of PPE will be assessed with a standardised three-grade system previously used in capecitabine clinical trials

SECONDARY OUTCOMES:
Change from Baseline EORTC QOLc30 at 3,4, 5,6 weeks | 3, 4,5 and 6 weeks
  The quality of life of the patients will be assessed with the EORTC QOLc30 module which has been developed and validated explicitly for patients suffering from cancer.
Change from Baseline Hand-foot syndrome 14 (HFS-14) at 3,4,5,6 weeks | 3, 4, 5 and 6 weeks
  this is a quality of life scale for patients experiencing radiation-induced PPE

OTHER OUTCOMES:
Change from Baseline Activities of daily living at 3,4,5,6 weeks | 3, 4, 5 and 6 weeks
  The ability of the patients to respond to their activities of daily living will be assessed with the Eastern Co-operative Oncology Group (ECOG)/WHO system
Treatment side-effects | During the 4 weeks
  The patients will report any possible side-effect due to the treatment (i.e rash)

CONTACTS AND LOCATIONS:
Locations (1):
- American Medical Centre, Nicosia, Cyprus

REFERENCES:
- [Derived] Stavrinou M, Tsitsi T, Astras G, Paikousis L, Charalambous A. A randomised controlled feasibility trial to evaluate Lawsonia inermis (henna)'s effect on palmar-plantar erythrodysesthesia induced by capecitabine or pegylated liposomal doxorubicin. Eur J Oncol Nurs. 2021 Apr;51:101908. doi: 10.1016/j.ejon.2021.101908. Epub 2021 Feb 15. PMID 33626423